CLINICAL TRIAL: NCT03295097
Title: A Prospective Multicenter Cohort Study to Evaluate The Characteristics and Clinical Implications of a Clinical Decision Support System and of Pharmacogenomic Information Relevant to Polypharmacy Actions in Patients With Advanced Illness Who Are Receiving Multiple Drugs for Pain and Other Disorders
Brief Title: Characteristics and Clinical Implications of a Clinical Decision Support System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospice of Henderson County, Inc. (Other)
Collaborators: Tabula Rasa HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TRHC2017-SERD101
Record Dates: First submitted 2017-08-23; First posted 2017-09-27 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2020-02

CONDITIONS: Chronic Illness; Opioid Use; Palliative Care
Keywords: pharmacogenomics
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Decision Support System (Other): The Clinical Decision Support System is composed of pharmacogenomic results and a pharmacist evaluated drug to drug interaction review. This system provides clinicians with patient-specific genetic information on opioid responsiveness and multi-drug interactions.
  Interventions: Other: Clinical Decision Support System

INTERVENTIONS:
Other: Clinical Decision Support System — The system provides clinicians with patient-specific genetic information on opioid responsiveness and multi-drug interactions. This clinical decision support system should improve the clinician's ability to identify the optimal pain medication and dosage, and reduce risks associated with multi-drug treatment.

SUMMARY:
The investigators propose to study the feasibility, acceptability, usability and outcomes of a new clinical decision support system for clinicians of opioid therapy in the context of specialist palliative care for serious chronic illness. The system provides clinicians with patient-specific genetic information on opioid responsiveness and multi-drug interactions. This clinical decision support system should improve the clinician's ability to identify the optimal pain medication and dosage, and reduce risks associated with multi-drug treatment. Investigators will conduct clinician survey's to collection information about the clinical decision support system. Investigators will also conduct patient related questionnaires to determine any benefits or improvements in quality of life and symptom management from the clinical decision support system.

ELIGIBILITY:
Inclusion Criteria:

Clinicians will be eligible if:

1. Physicians or nurse practitioners who are practicing hospice and palliative care
2. Responsible for making and implementing decisions about opioid therapy for pain

Patients will be identified by their treating clinicians. Patients will be eligible if:

1. > 18 years of age
2. Palliative Performance Score ≥ 30%
3. Reside in the community or at a nursing home
4. Have >1 serious chronic illness
5. Have an assessed life-expectancy of at least 4 weeks
6. Have a history of pain and have been taking prescribed opioid medication with a regimen that provides a minimum dose of 20 mg morphine or equivalent per day in scheduled doses for at least one week prior to recruitment
7. Is expected to continue opioid therapy for the duration of study participation
8. Is taking > 4 non-opioid medications, each in a regimen providing continuous treatment of pain or another disorder
9. Is expected to continue drug therapy for the duration of study participation
10. Able to read, understand, and provide Informed Consent to participate

Exclusion Criteria:

There are no exclusion criteria for clinicians.

Patients will be excluded if:

1. Pregnant women or women trying to become pregnant or nursing. Women of childbearing potential must use an acceptable method of birth control for the duration of the study. (acceptable forms are oral birth control pills, condoms in combination with spermicide foam, IUD, transdermal patches, birth control implants, vaginal ring)
2. Palliative Performance Score <30%
3. Have taken an investigational product in the last 30 days
4. Current use of illicit substances
5. Immediate family members of site staff, or site staff may not be enrolled in the study without first obtaining IRB authorization
6. Any other medical or physical abnormality, disease, or disorder that would prohibit the patient from completing study procedures in the judgement of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Clinician Feasibility | through study completion, an average of 24 months
  Clinical questionnaire to determine feasibility of the system
Clinician Usability | through study completion, an average of 24 months
  Clinical questionnaire to determine usability of the system

SECONDARY OUTCOMES:
Patient Quality of Life | through study completion,an average of 24 months
  Functional Assessment of Chronic Illness - Palliative (FACIT-PAL)
Patient Pain | through study completion, an average of 24 months
  Numerical Rating Scale to assess pain

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - MJHS Hospice and Palliative Care, New York, New York
  - Hospice of Henderson County, Inc. d/b/a Four Seasons Compassion for Life, Flat Rock, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided